CLINICAL TRIAL: NCT04054349
Title: The Effect of the Low Fodmap Diet on Gastrointestinal and Behavioral Problems in Children With Autism Spectrum Disorders
Brief Title: The Effect of the Low Fodmap Diet in Children With Autism Spectrum Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Marcia Nahikian-Nelms, Principal Investigator, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018H0543
Record Dates: First submitted 2019-08-07; First posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — FODMAP Diet

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low FODMAP Diet Group (Experimental): The parent/caregiver was given detailed nutrition education by the investigator concerning the low FODMAP diet and was asked to implement for 2 weeks.
  Interventions: Other: Low FODMAP diet
- Control Group (Habitual Diet) (No Intervention): The parent/caregiver was asked to continue their child's usual dietary intake for 2 weeks.

INTERVENTIONS:
Other: Low FODMAP diet — The low FODMAP diet group reduced the intake of FODMAP(fermentable oligosaccharides, disaccharides, monosaccharides, and polyols)
  Arms: Low FODMAP Diet Group

SUMMARY:
This study assesses the effect of the low fermentable oligosaccharides, disaccharides, monosaccharides, and polyols (FODMAP) diet on gastrointestinal (GI) and behavioral problems in children with autism spectrum disorder (ASD). The objectives of this study are: -To determine whether the low FODMAP diet causes a decrease in gastrointestinal problems related to ASD -To determine whether the low FODMAP diet causes a decrease in behavioral problems -To assess the effect of decreased gastrointestinal problems on reduction of behavioral problems

DETAILED DESCRIPTION:
In this study, participants were children with autism spectrum disorder (ASD) ages 6-17 years. Children with ASD were randomized to the low FODMAP diet or habitual diet for 2 weeks. At baseline and after a two-week intervention period, the parent/caregiver completed the Aberrant Behavior Checklist-Community and Pediatric Quality of Life Inventory Gastrointestinal Module. The parent/caregiver also completed a dietary food record, and stool consistency/frequency record (three days before start to intervention and the last three days of the intervention) of their children.

ELIGIBILITY:
Inclusion Criteria:

* 6-17 age range
* Diagnosed with autism spectrum disorder
* Parent/Caregiver report of constipation and /or abdominal pain. • ROME IV criteria was utilized to identify constipation (defined as the presence of two of more of the following symptoms: Two or fewer stools per week, at least 1 episode of fecal incontinence per week, history of retentive posturing or excessive volitional stool retention, history of painful or hard bowel movements, presence of a large fecal mass in the rectum, history of large diameter stools that can obstruct the toilet) • ROME IV criteria was utilized to identify abdominal pain (defined as the fulfilled at least 4 times per month and include all of the following: episodic or continuous abdominal pain that does not occur solely during physiologic events (eg, eating, menses), insufficient criteria for irritable bowel syndrome, functional dyspepsia, or abdominal migraine, the abdominal pain cannot be fully explained by another medical condition)

Exclusion Criteria:

* Under 6 and over 17 years old
* Having a specific restrictive diet to treat allergies or a specific chronic disease - Any history of abdominal surgeries
* Any history of chronic physiological GI disorders such as celiac, inflammatory bowel disease, eosinophilic esophagitis.
* Any chronic condition that may impact GI function such as thyroid disease, cystic fibrosis, or cardiac abnormalities

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Pediatric Quality of Life Inventory (PedsQL) Gastrointestinal Module-Parent Report | 2 weeks
  Before the study period and at the end of the two weeks, the effect of the low FODMAP diet on the severity of GI disorders was assessed with the Pediatric Quality of Life Inventory (PedsQL) Gastrointestinal Module-Parent Report. A 74-item survey with 14 scales items: stomach pain and hurt (6 items), discomfort when eating (5), food and drink limits (6), trouble swallowing (3), heartburn/reflux (4), nausea/vomiting (4), gas and bloating (7), constipation (14), blood in poop (2), diarrhea (7), worry about going poop (5), worry about stomachaches (2), medicines (4), and communication (5). Total Score: Sum of all the items over the number of items answered on all the Scales. Items are reverse-scored and transformed to a 0-100 scale so lower scores reflect worse GI dysfunction (As follows: 0=100, 1=75, 2=50, 3=25, 4=0). Response choices are in Likert-scale format ranging from 0 to 4 (0=Never, 1=Almost Never, 2=Sometimes, 3=Often, 4=Almost Always).

SECONDARY OUTCOMES:
Assessment of stool consistency | 2 weeks
  Consistency of the stool were recorded for 3 days before the study period and the last three days of the study using the Bristol stool scale. According to Bristol stool scale human stool is categorized into seven groups. Types 1 and 2 are defined as indications of constipation, Types 6 and 7 are indications of diarrhea, and Types 3, 4, and 5 show normal stool consistency. Daily stool consistency score was recorded. This was averaged and compared to the baseline and two weeks.
Assessment of stool frequency | 2 weeks
  Frequency of the stool were recorded for 3 days before the study period and the last three days of the study. Daily number of stools were recorded. This was averaged and compared to the baseline and two weeks.
Assessment of behavioral problems | 2 weeks
  Behavioral problems were determined before the study period and end of the study (after two weeks) using the Aberrant Behavior Checklist-Community (ABC-C). ABC-C checklist have 5 domains: 1) Irritability (includes agitation, aggression and self-injurious behaviors, 15 items); 2) Social Withdrawal (16 items); 3) Stereotypies (7 items); 4) Hyperactivity (16 items); and 5)Inappropriate Speech (4 items).The ABC-C is a 58-item questionnaire for caregivers/parent/caregivers and each item is scored as 0 (never a problem), 1 (slight problem), 2 (moderately serious problem), 3 (severe problem). it is not computed a total score based on the summation of all 58 items, as the subscales are largely independents. Higher scores indicate a higher severity of behavioral problems.
Energy and Nutrient Intake | 2 weeks
  The parent/caregiver recorded food consumption of children for three days before the study period and the last three days of the study.The data for the three day dietary record were entered into a computerized database. Energy, macronutrients and micronutrients were calculated using The Food Processor SQL - ESHA Research. 2006

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Nahikian-Nelms, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Nisonger Center, Columbus, Ohio, United States